CLINICAL TRIAL: NCT00986453
Title: A Prospective, Randomized, Controlled Study to Evaluate Use of the PEAK PlasmaBlade 4.0 in Bilateral Breast Reduction
Brief Title: PEAK PlasmaBlade 4.0 in Bilateral Breast Reduction
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00065
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Macromastia
Keywords: Breast Reduction; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Gigantomastia; Hyperthermia | interventions — Laser Therapy; Electrosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PlasmaBlade arm (Experimental): The PEAK PlasmaBlade will be used for the entirety of the breast reduction, including the skin incision.
  Interventions: Device: PEAK PlasmaBlade
- Standard of Care (Active Comparator): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Interventions: Procedure: Traditional Electrosurgery with scalpel

INTERVENTIONS:
Device: PEAK PlasmaBlade — The PEAK PlasmaBlade will be used for the entirety of the breast reduction, including the skin incision.
  Other Names: PlasmaBlade
  Arms: PlasmaBlade arm
Procedure: Traditional Electrosurgery with scalpel — Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Other Names: Scalpel; Electrosurgery; SOC
  Arms: Standard of Care

SUMMARY:
The objective of this clinical study is to evaluate the operative performance of the PEAK PlasmaBlade 4.0 during bilateral breast reduction; to monitor and record post-operative pain, adverse events and skin scarring following surgery; and compare these outcomes to the current standard of care (SOC).

DETAILED DESCRIPTION:
Bilateral breast reduction is a surgical procedure performed to remove excess breast tissue from both female breasts for therapeutic or cosmetic indications. The purpose of the breast reduction is to decrease the weight of the breasts and restructure the breast tissue for a more favorable appearance. Typically, a scalpel is used for the skin incision and a traditional electrosurgical device is used to cut away any excess tissue.

The PEAK PlasmaBlade™ uses pulsed radiofrequency (RF) energy and a highly-insulated handpiece design to enable precision cutting and coagulation at the point of application. The PlasmaBlade has received FDA clearance for use in plastic, general, and ear, nose, and throat (ENT) surgery, and has demonstrated a significantly reduced thermal injury profile in incised tissue compared to traditional electrosurgical devices. It is hypothesized that this benefit may improve the post-operative outcome of patients undergoing bilateral breast reduction.

A total of forty-five (45) subjects were enrolled into the study. Forty-three (43) underwent bilateral breast reduction, and two (2) subjects were withdrawn prior to surgery. Enrollment and surgeries took place between 18 September 2009 and 12 August 2011. Potential subjects were screened against the inclusion and exclusion criteria of the study protocol and were required to provide informed consent prior to enrollment. Following enrollment, subject operative sites were prospectively randomized to the SOC or PlasmaBlade (PB or PEAK) study groups and scheduled for bilateral breast reduction. Subjects were unaware of which device was used on which breast. Subjects were required to attend two follow-up visits after surgery, approximately one and six weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 60
2. Physically healthy, stable weight, non-smoker
3. Desiring bilateral breast reduction
4. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
5. Subject must be willing and able to comply with specified follow-up evaluations.
6. Female subjects must either be no longer capable of reproduction, or taking acceptable measures to prevent pregnancy during the study, and have a negative pregnancy test prior to participation in the study.

Exclusion Criteria:

1. Age younger than 20 or greater than 60 years old
2. Anticoagulation therapy which cannot be discontinued
3. Smoking (any kind)
4. Infection (local or systemic)
5. Cognitive impairment or mental illness
6. Severe cardiopulmonary deficiencies
7. Known coagulopathy
8. Immunocompromised
9. Prior history of breast cancer
10. Kidney disease (any type)
11. Currently taking any medication known to affect healing
12. Subjects who are status-post gastric banding or gastric bypass
13. Currently enrolled in another investigational device or drug trial
14. Unable to follow instructions or complete follow-up

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Gupta, MD, Principal Investigator — Gupta Plastic Surgery; Howard Rosenberg, MD, Principal Investigator — Accent on Aesthetics Plastic Surgery; Susan Downey, MD, Principal Investigator — Susan Downey, MD, FACS; Larry Pollack, MD, Principal Investigator — Del Mar Plastic Surgery; Hooman Soltanian, MD, Principal Investigator — University Hospital Cleveland
Locations (7):
- United States (7):
  - Providence St. Joseph's, Burbank, California
  - Verdugo Hills Hospital, Glendale, California
  - El Camino Hospital, Mountain View, California
  - Tri-City Medical Center, Oceanside, California
  - Sharp Outpatient Pavilion, San Diego, California
  - Rancho Bernardo Surgery Center, San Diego, California
  - University Hospitals, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects' individual breasts were prospectively randomized to the standard of care or PEAK PlasmaBlade.
Groups:
- Total Study Population: Subjects' individual breasts were prospectively randomized to the standard of care or PEAK PlasmaBlade.
Period: Overall Study
Arm/Group | Total Study Population
Started | 45
Completed | 43
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Study Population
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 41.12 (14.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: The difference in pain was measured by visual analog scale for 24 hours post-operatively and for 10 post-operative days twice daily between the SOC and PlasmaBlade operative sites.
  Wong-Baker FACES Visual Analog Scale, 0 (no hurt) to 10 (hurts worst). The results represent the mean of each subject's mean pain scores over 10 days.
Time Frame: 0 to 10 days postoperative
Population: Two subjects were removed from the analysis of secondary variables owing to protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: breasts
Groups:
- Standard of Care (SOC): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 43 | 43
Number analyzed (breasts) | 43 | 43
units on a scale | 4.47 (2.05) | 4.66 (2.08)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.4697, t-test, 2 sided

2. Secondary Outcome: Estimated Blood Loss
Time Frame: Intraoperative
Population: Two subjects were removed from the analysis of secondary variables owing to protocol deviations.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: breasts
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 43 | 43
Number analyzed (breasts) | 43 | 43
mL | 56.59 (48.44) | 64.27 (34.23)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.1470, t-test, 2 sided

3. Secondary Outcome: Operative Time
Time Frame: Intraoperative
Population: Two subjects were removed from the analysis of secondary variables owing to protocol deviations.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: breasts
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 43 | 43
Number analyzed (breasts) | 43 | 43
minutes | 37.40 (15.52) | 41.55 (11.61)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.0428, t-test, 2 sided

4. Secondary Outcome: Amount of Tissue Removed
Time Frame: Intraoperative
Population: Two subjects were removed from the analysis of secondary variables owing to protocol deviations.
Measure: Mean (Standard Deviation); unit: g
Units Other Than Participants: breasts
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 43 | 43
Number analyzed (breasts) | 43 | 43
g | 685.92 (347.08) | 649.18 (322.07)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.0776, t-test, 2 sided

5. Secondary Outcome: Dissection Performance
Description: Amount of tissue (g) removed over time (min)
Time Frame: Intraoperative
Population: Two subjects were removed from the analysis of secondary variables owing to protocol deviations.
Measure: Mean (Standard Deviation); unit: g/min
Units Other Than Participants: breasts
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 43 | 43
Number analyzed (breasts) | 43 | 43
g/min | 19.81 (10.65) | 15.99 (7.80)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/43
Other Adverse Events (participants affected / at risk) | 3/43 | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEAK PlasmaBlade (N=43) | Standard of Care (SOC) (N=43)
Hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — Second surgery was required to evacuate the hematoma.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEAK PlasmaBlade (N=43) | Standard of Care (SOC) (N=43)
Wound dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Surgical and medical procedures) | 1 (1) | 1 (1)
Seroma (Surgical and medical procedures) | 1 (1) | 3 (3) — One seroma could not be attributed to either device as the device identification field was not completed; therefore, 1 seroma was added to both groups in the tabulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less